CLINICAL TRIAL: NCT00907127
Title: Cardiac Autonomic Neuropathy in Patients With Metabolic Syndrome
Acronym: CAN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Associate Professor of Internal Medicine/MEND, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UM-5428; ADA
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic; Syndrome; CAN
MeSH Terms: conditions — Metabolic Syndrome; Syndrome | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mediterranean Diet and Exercise (Active Comparator): Mediterranean Diet and Exercise
  Interventions: Behavioral: Exercise and Diet (Metabolic Fitness Program)

INTERVENTIONS:
Behavioral: Exercise and Diet (Metabolic Fitness Program) — 6 month program of diet and exercise training and support.
  Other Names: Metabolic Fitness Program

SUMMARY:
The study will test whether damage of the heart nerves appears in patients before they develop diabetes.

DETAILED DESCRIPTION:
Patients who have mild abnormalities of blood sugar, high blood pressure, abnormal lipids and/or obesity can have a condition called metabolic syndrome. These patients are at high risk for diabetes and Cardiac Autonomic Neuropathy (CAN). Subjects with diagnosed metabolic syndrome will be expected to participate in the Metabolic Fitness Program which is a University of Michigan diet exercise program located in the Cardiology department at Domino Farms in Ann Arbor. Time required for this program and the study is 6 months. Clinic visits will involve Cardiac autonomic testing (CAN) procedures, PET scans and labs which will measure pre and post program intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have IGT or IFG and two other criteria of metabolic syndrome as defined by ATP III (IFG=fasting glucose ≥ 100 mg/dl (5.5 mmol/l))
2. Definition of IGT/IFG: IGT/IFG will be defined based on the ADA diagnostic guidelines following an oral glucose tolerance test (OGTT) [2].
3. Other Required Criteria (2 of the following):

   * Waist circumference ≥ 102 cm (40 inches) in men and ≥ 88 cm (35 inches) in women, {for Asian-Americans: men ≥ 88 cm (35 inches), women ≥ 78 cm (31 inches)}
   * Triglycerides ≥ 150 mg/dl (1.7 mmol/l) - patients on drug treatment with fibrates or nicotinic acid will be presumed to have triglycerides ≥ 150mg/dl and low HDL
   * HDL cholesterol < 40 mg/dl (1.0 mmol/l) in men and < 50 mg/dl (1.3 mmol/l) in women,
   * Blood pressure ≥ 130/≥ 85 mmHg
4. Age 18-65
5. Women of childbearing potential must be using contraception to prevent pregnancy

Exclusion Criteria:

1. Patients either pregnant or planning to become pregnant will be excluded

   * Women of childbearing potential will have a urine pregnancy test as part of the screening visit
   * Subjects who become pregnant during the study will undergo an exit visit and management of their IGT and Metabolic Syndrome will be returned to their primary care provider
2. Subjects with pre-existing cardiovascular disease including:

   * myocardial infarction
   * congestive heart failure
   * known arrhythmias
   * ventricular structural abnormalities and valvular disease
   * peripheral vascular disease
3. Subjects with hypoxemic lung or heart disease
4. Subjects with established diabetes
5. Laboratory evidence for a disease known to cause neuropathy within 3 months of screening will be an exclusion (those without known abnormality or those with a remote abnormality (> 3 months) will undergo the serologic screening)
6. Significant neurological disease (e.g., Parkinson's disease, epilepsy, recent stroke)
7. Subjects taking drugs which interfere with the uptake or metabolism of catecholamines
8. Subjects with known history of chronic kidney disease or who have significant hepatic disease (AST, ALT > 3 times upper limit for normal) or a history of previous kidney, pancreas or cardiac transplantation.
9. Subjects having taken systemic investigational drugs within the last 6 months
10. Inability or unwillingness of subject or legal guardian/representative to give written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic testing (CAN) | 6 months

SECONDARY OUTCOMES:
PET Scan | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Pop-Busui, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan Health System, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Mathew AV, Li L, Byun J, Guo Y, Michailidis G, Jaiswal M, Chen YE, Pop-Busui R, Pennathur S. Therapeutic Lifestyle Changes Improve HDL Function by Inhibiting Myeloperoxidase-Mediated Oxidation in Patients With Metabolic Syndrome. Diabetes Care. 2018 Nov;41(11):2431-2437. doi: 10.2337/dc18-0049. Epub 2018 Sep 10. PMID 30201848